CLINICAL TRIAL: NCT00079937
Title: A 1 Year, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Evaluation of Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Omalizumab in Children (6 - < 12 Years) With Moderate-severe, Persistent, Inadequately Controlled Allergic Asthma
Brief Title: Efficacy and Safety of Omalizumab in Children (6 - < 12 Years) With Moderate-severe, Inadequately Controlled Allergic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGE025AIA05
Record Dates: First submitted 2004-03-18; First posted 2004-03-22 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
Keywords: allergic; asthma; atopic; omalizumab; immunoglobulin E; IgE; anti-IgE
MeSH Terms: conditions — Asthma | interventions — Omalizumab; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Omalizumab (Experimental): Participants received omalizumab administered by subcutaneous injection every 2 or 4 weeks for a duration of 52 weeks. The omalizumab dose was based on the patient's body weight and total serum IgE level at Screening. The first 24 weeks of the treatment period was a fixed steroid phase where the steroid dose was maintained constant; in the following 28 weeks the steroid dose was adjustable, depending on the patient's condition. Following the 52-week treatment period, patients were followed up for an additional 16 weeks.
  Interventions: Drug: Omalizumab; Drug: Fluticasone
- Placebo (Placebo Comparator): Placebo was administered by subcutaneous injection every 2 or 4 weeks depending on the dosing schedule in the protocol for a total of 52 weeks. The first 24 weeks of the treatment period was a fixed steroid phase where the steroid dose was maintained constant; in the following 28 weeks the steroid dose was adjustable, depending on the patient's condition. Following the 52-week treatment period, patients were followed up for an additional 16 weeks.
  Interventions: Drug: Placebo; Drug: Fluticasone

INTERVENTIONS:
Drug: Omalizumab — The omalizumab dose administered, based on the patient's body weight and total serum IgE level at Screening, and the number of injections and injection volume was determined from the dosing tables in the protocol. Omalizumab 75 to 375 mg was administered subcutaneous (SC) every 2 or 4 weeks depending on the dose.
  Arms: Omalizumab
Drug: Placebo — Placebo was administered subcutaneous (SC) every 2 or 4 weeks depending on the dosing schedule in the protocol.
  Arms: Placebo
Drug: Fluticasone — Patients entered the study using their current formulation of any inhaled steroid (proprietary drug and device) ≥ 200 μg/day equivalent of fluticasone administered with a dry-powder inhaler.

SUMMARY:
A substance called immunoglobulin E (IgE), which is naturally produced by our body, has a key role in generating asthma attacks. In patients with allergies, there is an exaggerated production of IgE in response to specific substances such as pollens. Omalizumab is a new drug that inactivates IgE. This study tested the safety and efficacy of omalizumab against asthma attacks in children with allergic asthma.

DETAILED DESCRIPTION:
This study was designed to provide one year efficacy and safety data for subcutaneous (SC) omalizumab, compared to placebo in children (6 to < 12 years) with moderate to severe persistent asthma who have inadequate asthma control despite treatment according to National Heart, Lung and Blood Institute (NHLBI) step 3 or 4 (at least medium dose inhaled corticosteroids with or without other controller asthma medications).

ELIGIBILITY:
Inclusion criteria:

* Parent or legal guardian was informed of the study procedures and medications and gave written informed consent.
* Outpatient males and females aged 6 - < 12 years on study entry, with body weight between 20 and 150 kg.
* Total serum IgE level ≥ 30 to ≤ 1300 IU.
* Diagnosis of allergic asthma ≥ 1 year duration, according to American Thoracic Society (ATS) criteria, and a screening history consistent with clinical features of moderate or severe persistent asthma according to National Heart Lung and Blood Institute (NHLBI) guidelines.
* Positive prick skin test to at least one perennial allergen, documented within the past 2 years or taken at Screening. A radioallergosorbent test (RAST) could have been performed for patients with a borderline skin prick test result after consultation with Novartis clinical personnel.
* Patients with ≥ 12% increase in forced expiratory volume in 1 second (FEV1) over starting value within 30 minutes of taking up to 4 puffs (4x100 µg) salbutamol (albuterol) or nebulized salbutamol up to 5 mg (or equivalent of alternative B2-agonist) documented within the past year, at screening, during the run-in period, or prior to randomization. Patients were not to take their long acting B2-agonist (LABA) medication within 12 hours of reversibility testing.
* Clinical features of moderate or severe persistent asthma (at least step 3) despite therapy at step 3 or 4 (at least medium dose inhaled corticosteroid (ICS) - fluticasone dry-powder inhaler (DPI) ≥ 200 mg/day or equivalent with or without other controller medications).
* Documented history of experiencing asthma exacerbations and demonstrated inadequate symptom control during the last 4 weeks of run-in despite receiving an equivalent dose of fluticasone DPI ≥ 200 mg/day total daily ex-valve dose.

Exclusion criteria:

* Patients who received systemic corticosteroids for reasons other than asthma, beta-adrenergic antagonists by any route, anticholinergics within 24 hours of Screening, methotrexate, gold salts, cyclosporin or troleandomycin, or had received desensitization therapy with less than 3 months of stable maintenance doses prior to Screening.
* Patients with a history of food or drug related severe anaphylactoid or anaphylactic reaction, a history of allergy to antibiotics, with aspirin or other non-steroidal anti-inflammatory drugs (NSAID)-related asthma (unless the NSAID could be avoided), with active lung disease or acute sinusitis/chest infection, elevated serum IgE levels for other reasons, presence/history of a clinically significant uncontrolled systemic disease, cancer, abnormal, electrocardiogram (ECG) in the previous month, or platelets ≤ 100 x 109/L or clinically significant laboratory abnormalities at Screening.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 628 (Actual)
Dates: Start 2004-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- United States (56):
  - Alabama Allergy and Asthma Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Clinical Research Center, Little Rock, Arkansas
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - Pediatric Care and Medical Group, Huntington Beach, California
  - West Coast Clinical Trials, Long Beach, California
  - Southern California Research Center, Mission Viejo, California
  - Children's Hosptial of Orange County, Div Asthma, Allergy & Immunology, Orange, California
  - CA Allergy & Asthma Med Group, Palmdale, California
  - Dr. Joann Blessing-Moore, Palo Alto, California
  - Integrated Research Group, Riverside, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy and Asthma Medical Group & Research Center, San Diego, California
  - Allergy and Asthma Associates of Santa Clara Valley RC, San Jose, California
  - 1304 15th St, Santa Monica, California
  - Bensch Research Associates, Stockton, California
  - Allergy & Asthma Med Group of Diablo Valley CR, Walnut Creek, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Miami Children's Hospital, Miami, Florida
  - Georgia Pollens, Albany, Georgia
  - Family Allergy and Asthma Center, PC, Atlanta, Georgia
  - Aeroallergy Research Labs of Savannah, Inc, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Asthma & Allergy Center, Elliott, Maryland
  - Northeast Med Research Associates, North Dartmouth, Massachusetts
  - St. Louis University School of Medicine, St Louis, Missouri
  - Midwest Allergy & Asthma Clinic, Omaha, Nebraska
  - Ocean Allergy & Respiratory Research Center, Brick, New Jersey
  - UMDNJ, Newark, New Jersey
  - Womes And childrens Hospital of Buffalo, Buffalo, New York
  - Asthma & Allergy Associates, Ithaca, New York
  - Allergy and Asthma Diagnostic Office, Liverpool, New York
  - Island Medical Research (Allergy and Asthma Center), Rockville Centre, New York
  - Duke University Medical Center, Durham, North Carolina
  - Allergy & Asthma Center of North carolina, High Point, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Resp Dis of Children and Adolescents, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - 501 Howard Av, Altoona, Pennsylvania
  - West Penn Allegheny General Health System, Pittsburgh, Pennsylvania
  - Asthma and Allergy Associates, Upland, Pennsylvania
  - AAPRI Clinical Research Institute, Lincoln, Rhode Island
  - Allergy Assoc., The ASthma, Allergy & Sinus Ctr, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Pediatric Allergy/Immunology Associates, PA, Dallas, Texas
  - Pediatric Pulmonary Association of North Texas, Dallas, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - 7707 Fannin/Ste. 195, Houston, Texas
  - Sylvanna Research, San Antonio, Texas
  - Copperview Medical Center, South Jordan, Utah
  - Childrens Hospital of the Kings Daughters, Norfolk, Virginia
  - Virgina Commonwealth, Richmond, Virginia
  - A.S.T.H.M.A., Inc., Seattle, Washington
  - 508 W 6th Av, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fiocchi A, Chinthrajah RS, Ansotegui IJ, Sriaroon P, Mustafa SS, Raut P, Cameron B, Gupta S, Fleischer DM. Does Comorbid Food Allergy Affect Response to Omalizumab in Patients with Asthma? J Asthma Allergy. 2024 Sep 17;17:889-900. doi: 10.2147/JAA.S475517. eCollection 2024. PMID 39309477
- [Derived] Witonsky J, Elhawary JR, Millette LA, Holweg CTJ, Ko J, Raut P, Borrell LN. Similar response to omalizumab in children with allergic asthma from different racial backgrounds. J Allergy Clin Immunol Pract. 2023 Sep;11(9):2911-2913. doi: 10.1016/j.jaip.2023.03.055. Epub 2023 Apr 23. No abstract available. PMID 37088376
- [Derived] Busse WW, Szefler SJ, Haselkorn T, Iqbal A, Ortiz B, Lanier BQ, Chipps BE. Possible Protective Effect of Omalizumab on Lung Function Decline in Patients Experiencing Asthma Exacerbations. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1201-1211. doi: 10.1016/j.jaip.2020.10.027. Epub 2020 Oct 24. PMID 33223095
- [Derived] Szefler SJ, Casale TB, Haselkorn T, Yoo B, Ortiz B, Kattan M, Busse WW. Treatment Benefit with Omalizumab in Children by Indicators of Asthma Severity. J Allergy Clin Immunol Pract. 2020 Sep;8(8):2673-2680.e3. doi: 10.1016/j.jaip.2020.03.033. Epub 2020 Apr 13. PMID 32298853
- [Derived] Lanier B, Bridges T, Kulus M, Taylor AF, Berhane I, Vidaurre CF. Omalizumab for the treatment of exacerbations in children with inadequately controlled allergic (IgE-mediated) asthma. J Allergy Clin Immunol. 2009 Dec;124(6):1210-6. doi: 10.1016/j.jaci.2009.09.021. PMID 19910033

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 421 | 207
Completed | 352 | 175
Not Completed | 69 | 32
Not completed — Adverse Event | 2 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 2
Not completed — Subject no longer requires study drug | 3 | 0
Not completed — Protocol Violation | 8 | 6
Not completed — Withdrawal by Subject | 21 | 7
Not completed — Lost to Follow-up | 12 | 5
Not completed — Administrative problems | 22 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 421 | 207 | 628
Age Continuous [Mean (Standard Deviation); unit: years] | 8.7 (1.7) | 8.4 (1.7) | 8.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 69 | 203
  Male | 287 | 138 | 425
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 69 | 30 | 99
  White | 249 | 128 | 377
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 103 | 47 | 150

OUTCOME MEASURES:

1. Secondary Outcome: Change in Mean Nocturnal Asthma Symptom Score From Baseline to the End (Last 4 Weeks) of the 24-week Fixed-dose Steroid Treatment Period
Description: Nocturnal asthma symptom was measured daily on a scale of 0 to 4 in response to the question "How did you sleep last night?", with 0 as the best response and 4 as the worst response. The mean of the last 4 weeks of the 24-week fixed-dose steroid treatment period was calculated; for patients who discontinued prematurely, the mean of the last 28 days before discontinuation was calculated. A negative change in mean score indicated improvement.
Time Frame: Baseline to the end (last 4 weeks) of the 24-week fixed-dose steroid treatment period
Population: Modified intent-to-treat population: All patients who were randomized, excluding patients from 2 sites due to Good Clinical Practice non-compliance. Excluded patients were replaced with patients at other sites to maintain statistical power.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 382 | 191
Units on a scale | -0.63 (0.72) | -0.50 (0.71)

2. Primary Outcome: Rate of Clinically Significant Asthma Exacerbations Per Patient in the 24-week Fixed-dose Steroid Treatment Period
Description: A clinically significant asthma exacerbation was defined as a worsening of asthma symptoms, as judged clinically by the investigator, requiring doubling of the baseline inhaled corticosteroid dose and/or treatment with systemic rescue corticosteroids for at least 3 days. The exacerbations rate per patient was derived using Poisson model adjusted by time at risk and the following covariates: country, exacerbation history, and dose schedule. A patient's person-days at risk was taken as the total amount of time (in days) he/she spent in the 24-week fixed-dose steroid treatment period.
Time Frame: Baseline to end of the fixed-dose steroid treatment period (Week 24)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Exacerbations per patient per 24-weeks
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 384 | 192
Exacerbations per patient per 24-weeks | 0.45 [0.36 to 0.55] | 0.64 [0.49 to 0.83]

3. Secondary Outcome: Rate of Clinically Significant Asthma Exacerbations Per Patient in the 52-week Treatment Period
Description: A clinically significant asthma exacerbation was defined as a worsening of asthma symptoms, as judged clinically by the investigator, requiring doubling of the baseline inhaled corticosteroid dose and/or treatment with systemic rescue corticosteroids for at least 3 days. The exacerbations rate per patient was derived using Poisson model adjusted by time at risk and the following covariates: country, exacerbation history, and dose schedule. A patient's person-days at risk was taken as the total amount of time (in days) he/she spent in the 52-week treatment period.
Time Frame: Baseline to end of the treatment period (Week 52)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Exacerbations per patient per year
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 384 | 192
Exacerbations per patient per year | 0.78 [0.65 to 0.94] | 1.36 [0.92 to 1.71]

4. Secondary Outcome: Change in Mean Daily Number of Puffs of Asthma Rescue Medication From Baseline to the End (Last 4 Weeks) of the 24-week Fixed-dose Steroid Treatment Period
Description: Patients were instructed to record the number of puffs of rescue medication they took twice daily in a diary. The mean daily number of puffs during the last 4 weeks of the 24-week fixed-dose steroid treatment period was calculated; for patients who discontinued prematurely, the mean of the last 28 days before discontinuation was calculated. A negative change in mean daily number of puffs indicated reduced use of rescue medication.
Time Frame: Baseline to the end (last 4 weeks) of the 24-week fixed-dose steroid treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Puffs
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 381 | 191
Puffs | -1.3 (2.84) | -1.0 (2.50)

5. Secondary Outcome: Change in Pediatric Asthma Quality of Life Questionnaire (Standardized) [PAQLQ(S)] Scores From Baseline to the End of the 24-week Fixed-dose Steroid Treatment Period (Week 24)
Description: PAQLQ measures functional problems that are most troublesome to children with asthma. PAQLQ has 23 questions in 3 domains (activity limitation=5, emotional function=8, symptoms=10). Patients responded to each question on a 7-point Likert scale. Overall PAQLQ score is mean of 23 questions; each domain score is mean of questions in that domain. Minimum possible value is 1 (maximum impairment); maximum possible value is 7 (no impairment). Positive change indicated improvement. The analysis included country, baseline PAQLQ value, and dosing schedule (2-weekly/4-weekly) as factors and covariates.
Time Frame: Baseline to the end of the 24-week fixed-dose steroid treatment period (Week 24)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 375 | 187
Units on a scale
  Activity limitation | 0.85 [0.72 to 0.99] | 0.76 [0.59 to 0.93]
  Emotional function | 0.89 [0.76 to 1.03] | 0.91 [0.74 to 1.09]
  Symptoms | 0.99 [0.85 to 1.13] | 0.93 [0.76 to 1.10]
  Overall (total) | 0.92 [0.80 to 1.05] | 0.89 [0.73 to 1.05]

6. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event
Description: See Adverse Events module for details.
Time Frame: Baseline to end of the study (Week 68)
Population: Safety population: All patients who received any study drug and had at least 1 post-baseline safety assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 421 | 207
Percentage of participants | 90.3 | 93.7

ADVERSE EVENTS:
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 27/421 | 26/207
Other Adverse Events (participants affected / at risk) | 374/421 | 194/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=421) | Placebo (N=207)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 6
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Tic (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=421) | Placebo (N=207)
Abdominal pain (Gastrointestinal disorders) | 23 | 12
Diarrhoea (Gastrointestinal disorders) | 20 | 12
Vomiting (Gastrointestinal disorders) | 34 | 24
Pyrexia (General disorders) | 59 | 20
Bronchitis (Infections and infestations) | 36 | 29
Ear infection (Infections and infestations) | 22 | 11
Gastroenteritis (Infections and infestations) | 19 | 15
Gastroenteritis viral (Infections and infestations) | 23 | 7
Influenza (Infections and infestations) | 51 | 28
Nasopharyngitis (Infections and infestations) | 117 | 56
Pharyngitis (Infections and infestations) | 36 | 18
Pharyngitis streptococcal (Infections and infestations) | 19 | 13
Rhinitis (Infections and infestations) | 25 | 20
Sinusitis (Infections and infestations) | 70 | 38
Tonsillitis (Infections and infestations) | 7 | 11
Upper respiratory tract infection (Infections and infestations) | 68 | 46
Viral upper respiratory tract infection (Infections and infestations) | 34 | 26
Headache (Nervous system disorders) | 58 | 33
Asthma (Respiratory, thoracic and mediastinal disorders) | 290 | 170
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 25
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 33 | 16
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 35 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.